CLINICAL TRIAL: NCT03664791
Title: Prospective, Multicentre Evaluation of the Vanguard Rocc Rotating Platform Knee Prosthesis - Clinical and Radiographic Outcomes
Brief Title: Vanguard Rocc Post Market Surveillance
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: BMETEU.CR.EU32
Record Dates: First submitted 2018-09-06; First posted 2018-09-11 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2023-06

CONDITIONS: Osteoarthritis, Knee; Rheumatoid Arthritis; Traumatic Arthritis; Posttraumatic Deformity; Varus Deformity; Valgus Deformity; Osteotomy; Arthrodesis
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis, Rheumatoid; Ankylosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Vanguard Rocc knee implant: Patient in need for a total knee arthroplasty and who met the inclusion/ exclusion criteria and received the Vanguard Rocc implant
  Interventions: Procedure: Vanguard Rocc

INTERVENTIONS:
Procedure: Vanguard Rocc — Patient operated with the Vanguard Rocc knee prosthesis

SUMMARY:
The objective of this project is to obtain prospective, multi-center, long term (10 year) clinical data on the Vanguard Rocc knee prosthesis. Patient and knee function will be collected along with knee stability, the knee motion, functional recuperation, radiographic and survivorship data.

DETAILED DESCRIPTION:
The Vanguard rotating platform knee prosthesis (Vanguard ROCC) was launched in March 2009. Therefore there is a need to show the safety and performance of the Vanguard ROCC at long term.

A maximum of 10 sites will be involved in this study. This number of clinical centers will permit assessment of consistency among a multitude of investigators.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria should be in accordance with Indications for Use for Vanguard-ROCC® Knee

System specifically:

* Painful and disabled knee joint resulting from osteoarthritis, rheumatoid arthritis, traumatic arthritis where one or more compartments are involved.
* Correction of varus, valgus, or posttraumatic deformity.
* Correction or revision of unsuccessful osteotomy, or arthrodesis.

Additional inclusion criteria include:

* Male or female.
* 18 years of age or older
* Subjects willing to return for follow-up evaluations

Exclusion Criteria:

Exclusion criteria should be in accordance with Absolute and Relative Contraindications for Use for Vanguard-ROCC Knee system: Absolute contraindications include: infection, sepsis, osteomyelitis, and failure of a previous joint replacement.

Relative contraindications include:

* Uncooperative patient or patient with neurologic disorders who are incapable of following directions,
* Osteoporosis,
* Metabolic disorders which may impair bone formation,
* Osteomalacia,
* Distant foci of infections which may spread to the implant site,
* Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram,
* Vascular insufficiency, muscular atrophy, neuromuscular disease,
* Incomplete or deficient soft tissue surrounding the knee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in need of a total knee arthroplasty which receive the Vanguard Rocc knee device and who meet all of the inclusion and none of the exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2009-10-23 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional outcomes assessment | 10 years
  The American Knee Society Clinical Rating System (original method) : Evaluation of the knee joint and functional assessment of patients.
  Subscale knee assessment: judgement of pain (50 points), stability (25 points)and range of motion (25 points (5 degrees is 1 point). Flexion contracture, extension lag and malalignment should be dealt with as deductions. Maximum Knee score of 100 points.
  Subscale functional assessment: assessment of patient function for walking distance (50 points)and stair climbing (50points), with deductions for walking aids. Maximum Function score is 100 points.

SECONDARY OUTCOMES:
Radiographic outcomes assessment | 10 years
  The Knee Society Total Knee Arthroplasty Roentgenographic Evaluation and Scoring System by Ewald: radiographic assessment for component position, leg and knee alignment, and the prosthesis-bone interface or fixation.
  To assess the quality of the fixation: the prosthetic interface has a numerical score for components femur, tibia and patella.
  The scoring system for each of the three components is determined by measuring the width of the radiolucent lines for each of the zones in millimeters for each of the three components. The total widths are added for each zone for each of the three components. This total produces a numerical score for each component.
  Example for interpretation for a seven-zone tibial component: 4 or less and nonprogressive is not significant; 5-9 should be closely followed for progression; and 10 or greater signifies possible or impending failure regardless of symptoms.
Assesment of health-related quality of life using the EQ-5D score | 10 years
  Euroqol-5 dimensions by the EuroQol Group (EQ-5D) consists of a descriptive system of health-related quality of life by a questionnaire and a thermometer scale. The Questionnaire comprises five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) with each 5 levels: no problems (level 1), slight problems (level 2), moderate problems, (level 3) severe problems (level 4) and extreme problems (level 5). The digits for the five dimensions can be combined into a 5-digit number and may be converted to a score (maximum is 1), defined by the health state classification.
  The Thermometer generates a self rating of current health-related quality of life and has end points of 100 (best imaginable health state) at the top, and 0 (worst imaginable health state) at the bottom. It should be used with the 5-digit health state classification to build a composite picture of the respondent's health status.
Safety and performance of the device by recording all adverse events | 10 years
  assessment of all occured adverse events
Calculation of survivorship using revision of prosthesis as the failure event | 10 years
  survivorship calculation by Kaplan-Meier technology

CONTACTS AND LOCATIONS:
Overall Officials: Paola Vivoda, Study Director — Zimmer Biomet
Locations (9):
- ZNA Jan Palfijn, Merksem, Belgium
- Denmark (2):
  - Sydvestjysk Hospital, Grindsted
  - Hvidovre University Hospital, Hvidovre
- France (5):
  - Clinique Pasteur, Guilherand-Granges
  - Clinique des Fontaines, Melun
  - Clinique d'Argonayy, Pringy
  - Clinique d'Argonay, Pringy
  - Clinique du Renaison, Roanne
- South West London Elective Orthopaedic centre - EPSOM General Hospital, Epsom, United Kingdom